CLINICAL TRIAL: NCT06684470
Title: Novel Pilot Study to Treat Symptoms of IBS With Diarrhea Using Combination Therapy of a Low-FODMAP Diet and a Neuromodulator
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Lacy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-011874
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: IBS - Irritable Bowel Syndrome; Diarrhea
Keywords: Diarrhea; IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirtazapine Group (Experimental): Subjects will present at Mayo Clinic through a doctor's appointment and a diagnosis of irritable bowel syndrome will be receiving mirtazapine by pill form.
  Interventions: Drug: Mirtazapine
- Placebo Group (Placebo Comparator): Subjects will present at Mayo Clinic through a doctor's appointment and a diagnosis of irritable bowel syndrome will be receiving placebo by pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mirtazapine — mirtazapine will be told to use 1 pill 1 hour before bedtime for the first week (7.5 mg po q.h.s.), 2 pills before bedtime during the second week of therapy (15 mg po q.h.s.), 3 pills (22.5 mg po q.h.s.) 1 hour before bedtime for the third week, and 4 pills (30 mg po q.h.s.) 1 hour prior to bedtime for the remainder of the study.
  Other Names: Remeron
  Arms: Mirtazapine Group
Other: Placebo — Placebo will be told to use 1 pill 1 hour before bedtime for the first week (7.5 mg po q.h.s.), 2 pills before bedtime during the second week of therapy (15 mg po q.h.s.), 3 pills (22.5 mg po q.h.s.) 1 hour before bedtime for the third week, and 4 pills (30 mg po q.h.s.) 1 hour prior to bedtime for the remainder of the study.
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to study the added benefit of treating IBS symptoms with a medication called mirtazapine in treating IBS symptoms when paired with a low-FODMAP diet compared to a low-FODMAP diet alone. FODMAP stands for fermentable oligosaccharides, disaccharides, monosaccharides, and polyols. These are short-chain carbohydrates that can cause digestive distress in some people.

You have been asked to take part in this research because you have symptoms of diarrhea-predominant irritable bowel syndrome that may respond to treatment with a combination of a medication called mirtazapine and a low-FODMAP diet.

DETAILED DESCRIPTION:
We hypothesize that adult patients with IBS-D treated with a combination of a low FODMAP diet and mirtazapine will have a greater improvement in global IBS symptoms including abdominal pain and diarrhea in addition to improved quality of life compared to those treated with a low-FODMAP diet only. Global improvement in IBS symptoms will be evaluated using the validated IBS-SSS questionnaire. We will evaluate changes in quality of life using a validated IBS-QoL questionnaire. We will assess the improvement in abdominal pain using a numerical rating system and assess improvements in diarrhea using the Bristol stool form scale. We will assess responses to bloating using a Mayo bloating questionnaire forms. We will assess improvement in diarrhea using the Bristol stool form scale.

Improvement in anxiety and any other descriptive information as provided by patients including patients reporting impression of overall severity of symptoms at the beginning, middle, and end of study.

Irritable bowel syndrome (IBS) is a common gastrointestinal (GI) disorder that affects up to 10% of the United States adult population. IBS is characterized by recurrent abdominal pain and altered bowel habits, diagnosed using the Rome IV criteria. Approximately one-third of all IBS patients are classified as having IBS with diarrhea (IBS-D), which has no validated treatment algorithm. The American College of Gastroenterology IBS guideline recommends the low-FODMAP (fermentable oligo-, di-, monosaccharide, and polyol) diet as a safe and modestly effective treatment. An analysis of 7 randomized, controlled trials found that the low-FODMAP diet was associated with an improvement in global IBS symptoms. However, despite following the low-FODMAP diet, many patients have persistent abdominal pain, which can be difficult to treat. The mechanisms underlying chronic abdominal pain in patients with IBS are unknown, although visceral and central hypersensitivity are thought to play a role. No medication is FDA-approved for the treatment of abdominal pain in IBS. Mirtazapine is an atypical antidepressant that acts on several classes of receptors. In a small open-label study mirtazapine improved IBS-D symptoms, including abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the inclusion criteria to participate in this study:

  * Adults (ages 18-70)
  * Score of >175 on the IBS-SSS questionnaire
  * Must meet Rome IV criteria for IBS-D
  * If subject is of reproductive capability a negative urine pregnancy test must be available prior to entering the study
  * Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* All candidates meeting any of the below exclusion criteria at baseline will be excluded from study participation:

  * Score of < 175 on the IBS-SSS
  * Prior diagnoses of: known celiac disease, small intestinal bacterial overgrowth, inflammatory bowel disease, or microscopic colitis
  * Ongoing significant anxiety or depression
  * A history of a known side effect to mirtazapine
  * Prior treatment with a low FODMAP diet or mirtazapine without clinical benefit
  * Active alcohol or drug abuse
  * Inability to read or understand the consent form
  * Any other medical or psychological reason that would prevent active participation in a research study
  * Pregnant females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Resolution of Irritable Bowel Syndrome | 49 days
  Evaluate global improvement in IBS symptoms using the validated IBS-SSS
Abdominal Pain Score | 49 days
  Assess improvement in abdominal pain using a numerical rating system
Stool Form Scale | 49 days
  Assess improvement in diarrhea using the Bristol stool form scale
Mayo Bloating Scale | 49 days
  Assess response to bloating using a validated Mayo bloating questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Lacy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No